CLINICAL TRIAL: NCT06679842
Title: Early Ascitis Parencentesis at Day-1 to Assess Antibiotic Response in Spontaneous Bacterial Peritonitis
Brief Title: Early Ascitis Parencentesis in SBP
Acronym: PAPISLA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024/901
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Cirrhosis; Spontaneous Bacterial Peritonitis
Keywords: resistant bacteria; spontaneous bacterial peritonitis; antibiotic; early paracentesis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one arm (Experimental)
  Interventions: Diagnostic Test: ascitis paracentesis

INTERVENTIONS:
Diagnostic Test: ascitis paracentesis — ascitis paracentesis

SUMMARY:
Paracentesis at 48 hours, as recommended in international guidelines, could delay the time to effective antibiotic therapy in cases of SBP with germs resistant to empirical antibiotic therapy. Earlier paracentesis at 24 hours could save time in initiating the right antibiotic therapy and improve prognosis.

DETAILED DESCRIPTION:
International recommendations call for exploratory paracentesis to be performed on admission in all cirrhotic patients presenting with clinical ascites. Based on data from a study published in 1990, the diagnosis of spontaneous bacterial infection (SBP) is defined by the presence of neutrophils (PNN) ≥ 250/mm3 in ascites fluid, irrespective of the bacteriological culture result . Although culture of ascites fluid is negative in 40-60% of confirmed cases of ISLA, and it takes 2-5 days to obtain a result, it remains essential to best adapt antibiotic therapy. Empirical antibiotic therapy is started as soon as SBP is diagnosed. Response to antibiotic therapy is defined as a reduction of more than 25% in the number of PNN in ascites sampled 48 hours after initiation of treatment. However, the landmark study by Akriviadis et al showed that the mean number of PNN fell significantly as early as 24 hours after the start of treatment, with a drop in PNN as early as the 6th hour. In the absence of a response to treatment, antibiotic therapy should be modified on the basis of culture results if positive, or empirically in the absence of bacteriological documentation. A recent study showed that a reduction in the number of PNN in ascites fluid after effective empirical antibiotic therapy was significantly associated with improved survival. Thus, waiting 48 hours to perform a follow-up paracentesis could delay the adjustment of effective antibiotic therapy in the event of initial non-response, and thus worsen the prognosis of SBP.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or over
* Affiliation with a French social security
* Signature of the informed consent form
* Cirrhosis
* Ascites fluid infection with PNN > 250/mm3

Exclusion Criteria:

* Pregnant women
* Persons deprived of their liberty by judicial or administrative decision; persons under psychiatric care.
* Adults under legal protection
* Subjects within the exclusion period of another study
* Other cause of abdominal infection than SBP
* Intra-abdominal surgery < 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-11 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the percentage drop in neutrophils in ascites on Day 1 | 24 hours
  Evaluate the percentage drop in neutrophils in ascites on Day 1, in order to assess the best threshold for predicting response to antibiotic therapy on Day 1 (judged on Day 2) in patients with ascites fluid infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatology Unit, CHU Besancon, Besançon, Doubs, France

IPD SHARING:
Plan to Share IPD: No